CLINICAL TRIAL: NCT07327515
Title: A Phase I/II Study of PET/CT-Guided Biological Target Volume Delineation and Dose Optimization for Radioactive Seed Implantation Therapy in Malignant Tumors
Brief Title: PET/CT-Guided Biological Target Volume Delineation and Dose Optimization for Radioactive Seed Implantation Therapy in Malignant Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Li Min (Other)
Responsible Party: Sponsor-Investigator, Li Min, Vice Director, Jinan Military General Hospital
Organization: Jinan Military General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 960HP20251026
Record Dates: First submitted 2025-11-16; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Malignant Tumors
Keywords: PET/CT-Guided Brachytherapy; Iodine-125 Seed Implantation; Molecular Imaging-Guided Therapy; Biology-Guided Dose Planning
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are assigned in parallel to three groups: CT-guided, PET/CT-guided standard dose, and PET/CT-guided biological dose optimization. Exploratory cohorts may use tumor-specific PET tracers, including PSMA, FAPI, and other emerging agents, to refine biological targeting and predictive modeling.
Who Masked: Outcomes Assessor
Masking Description: Due to the procedural nature of seed implantation, participants and treating clinicians cannot be blinded. However, independent radiologists and nuclear medicine physicians who evaluate imaging outcomes (e.g., tumor response, PET metabolic parameters, local control) will be blinded to group allocation and treatment details. Blinded image review will include: (1) PET/CT parameter assessment (SUVmax, MTV, TLG), (2) Radiographic response evaluation (RECIST 1.1 criteria), (3) Dosimetric verification (D90, V100, V150). All imaging data will be anonymized before evaluation to minimize potential bias in efficacy and dosimetric assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CT-Guided Radioactive Seed Implantation (Active Comparator): CT-guided 125I seed brachytherapy with a standard dose prescription. Target delineation based on contrast-enhanced CT. Post-implant dosimetry will verify D90, V100, V150, and organ-at-risk constraints.
  Interventions: Procedure: CT-Guided Radioactive Seed Implantation
- PET/CT-Guided Radioactive Seed Implantation - Standard Dose (Experimental): PET/CT-guided 125I seed implantation using PET/CT to support anatomical target delineation without SUV-based biological sub-volume definition. A standard uniform-dose prescription is applied. Post-implant dosimetry verifies target coverage and organ-at-risk constraints.
  Interventions: Procedure: PET/CT-Guided Radioactive Seed Implantation
- PET/CT-Guided Radioactive Seed Implantation - Biological Dose Optimization (Experimental): PET/CT-guided 125I seed implantation incorporating SUV-based biological sub-volume identification. High-SUV regions receive selective dose escalation through adjustments in seed activity or spatial seed distribution while maintaining organ-at-risk constraints.
  Interventions: Procedure: PET/CT-Guided Radioactive Seed Implantation (Biological Dose Optimization)
- Specific PET/CT-Guided Radioactive Seed Implantation (PSMA/FAPI Subgroup) (Experimental): Tumor-specific PET tracers such as PSMA and FAPI are used in selected subgroups to enhance lesion visualization and biological characterization for planning 125I seed implantation. Additional tracers are not currently in clinical use within the department but may be incorporated in future protocol amendments as availability allows.
  Interventions: Procedure: Tumor-Specific PET/CT-Guided Radioactive Seed Implantation (PSMA/FAPI Subgroup)

INTERVENTIONS:
Procedure: CT-Guided Radioactive Seed Implantation — CT-guided implantation of 125I radioactive seeds for localized treatment of malignant tumors. The target area is delineated on contrast-enhanced CT images, and seeds are implanted according to a treatment planning system (TPS) with a prescribed dose of about 100 Gy. Post-procedure dosimetry will confirm D90, V100, and V150, as well as organ-at-risk (OAR) dose constraints.
  Arms: CT-Guided Radioactive Seed Implantation
Procedure: PET/CT-Guided Radioactive Seed Implantation — PET/CT-guided 125I seed implantation performed using PET/CT fusion to support anatomical target delineation without SUV-based biological sub-volume definition. A standard uniform-dose treatment plan is implemented, and post-implant dosimetric evaluation is used to confirm target coverage and compliance with organ-at-risk constraints.
  Arms: PET/CT-Guided Radioactive Seed Implantation - Standard Dose
Procedure: PET/CT-Guided Radioactive Seed Implantation (Biological Dose Optimization) — PET/CT-guided 125I seed implantation for the treatment of malignant tumors. The biological target volume (BTV) is defined using 18F-FDG PET/CT fused with planning CT to improve target accuracy and tumor coverage. The prescribed dose is approximately 100 Gy. Post-implant verification includes D90, V100, and OAR constraints.
  Arms: PET/CT-Guided Radioactive Seed Implantation - Biological Dose Optimization
Procedure: Tumor-Specific PET/CT-Guided Radioactive Seed Implantation (PSMA/FAPI Subgroup) — 125I seed brachytherapy guided by tumor-specific PET/CT imaging. Tracers such as PSMA (for prostate cancer) and FAPI (for pancreatic, colorectal, and fibrotic tumors) identify biologically active regions for targeted dose escalation. High-uptake areas (SUVmax > threshold determined by tracer characteristics) receive escalated doses of approximately 120-150 Gy through increased seed density or activity, while normal tissues remain within tolerance limits.
  Arms: Specific PET/CT-Guided Radioactive Seed Implantation (PSMA/FAPI Subgroup)

SUMMARY:
This prospective, open-label Phase I/II trial evaluates a PET/CT-guided planning strategy for radioactive seed implantation therapy in malignant solid tumors. The approach integrates metabolic information from PET/CT into brachytherapy planning to improve the accuracy of biological target volume delineation, enhance dose coverage, and support biologically informed dose delivery. Eligible participants are assigned to one of three arms: conventional CT-guided implantation, PET/CT-guided standard-dose implantation, or PET/CT-guided biologically optimized implantation. All participants undergo image-guided treatment followed by post-implant dosimetric verification and standardized clinical follow-up.

Primary endpoints include technical success rate, dosimetric superiority, and 6-month local control. Secondary endpoints include dosimetric indices (D90, V100, conformity index, homogeneity index), pain relief, quality of life (EORTC QLQ-C30), treatment-related adverse events (CTCAE v5.0), progression-free survival (PFS), failure-free survival (FFS), and overall survival (OS). Exploratory analyses will evaluate associations between baseline PET metabolic parameters (SUVmax, metabolic tumor volume) and clinical outcomes, assess the feasibility of SUV-guided dose painting, and compare the performance of tumor-specific tracers (such as PSMA and FAPI) with FDG for target delineation and treatment response prediction.

The central hypothesis is that PET/CT-guided planning-particularly when incorporating biological dose optimization-will achieve superior dosimetric performance and improved local control and survival outcomes compared with conventional CT-guided implantation.

DETAILED DESCRIPTION:
This prospective, open-label Phase I/II trial evaluates a molecular-imaging-guided optimization strategy that integrates PET/CT into radioactive seed implantation therapy to improve target delineation accuracy, biological precision, and therapeutic efficacy in malignant solid tumors. Conventional CT-guided planning relies primarily on anatomical visualization and geometric dose coverage but does not incorporate intratumoral biological heterogeneity, which may result in uneven dose distribution and increased risk of local recurrence. To address this limitation, the trial incorporates PET/CT-based biological target volume (BTV) delineation and standardized uptake value (SUV)-driven dose modulation to achieve individualized, biologically optimized treatment planning.

Eligible participants with measurable solid tumors suitable for percutaneous implantation are assigned to one of three groups: (1) conventional CT-guided implantation, (2) PET/CT-guided implantation with standard dosing, and (3) PET/CT-guided implantation with biological dose optimization based on metabolic activity quantified by SUV measures. PET/CT is used to identify metabolically active sub-volumes for selective dose escalation while sparing normal tissues, achieved by adjusting seed activity or spatial distribution to deliver intensified irradiation to high-SUV tumor regions. In addition to standard 18F-FDG PET/CT, tumor-specific tracers are evaluated in selected subgroups to enhance lesion visualization and biological characterization, including 18F-PSMA for prostate cancer, 68Ga-FAPI for pancreatic, colorectal, and fibrotic tumors, 18F-FES for ER-positive breast cancer, and 18F-FMISO or 18F-FAZA for hypoxia detection and targeted dose escalation.

Primary endpoints include technical success rate, dosimetric superiority, and 6-month local control defined by imaging and clinical criteria. Secondary endpoints include dosimetric parameters (D90, V100, conformity index, homogeneity index), pain relief, quality of life (EORTC QLQ-C30), treatment-related adverse events (CTCAE v5.0), and time-to-event outcomes including progression-free survival (PFS), failure-free survival (FFS), and overall survival (OS). Exploratory analyses evaluate correlations between baseline PET parameters (SUVmax, metabolic tumor volume, total lesion glycolysis), radiomics features, and clinical outcomes, as well as early metabolic response (ΔSUVmax at 4-6 weeks) as a predictor of local control.

The central hypothesis is that PET/CT-guided biological optimization will enhance dosimetric conformity, improve local tumor control and survival outcomes, reduce recurrence, and contribute to better symptom relief and quality-of-life measures. Overall, the trial aims to establish a personalized, molecular-imaging-based framework for radioactive seed implantation therapy in malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Pathologically or clinically confirmed malignant tumor (solid tumor, lymphoma, or leukemia with a localized lesion suitable for radioactive seed implantation).
3. Tumor site accessible for image-guided implantation, with a target lesion visible on CT or PET/CT.
4. Life expectancy of at least 6 months.
5. Ability to undergo PET/CT imaging (FDG or tumor-specific tracers such as PSMA or FAPI).
6. Signed written informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Uncontrolled infection or active systemic inflammatory disease.
3. Severe cardiopulmonary dysfunction that contraindicates interventional procedures (e.g., heart failure, severe COPD).
4. Coagulation disorders (INR > 1.5 or platelet count < 50 × 10⁹/L).
5. Known allergy or intolerance to radiopharmaceuticals or iodinated contrast media.
6. Prior radiation therapy overlapping with the planned implantation area.
7. Participation in another clinical trial within the past 30 days that may interfere with study results.
8. Any medical or psychosocial condition considered unsuitable for study participation by the investigators (e.g., poor compliance, unstable clinical status).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success Rate | Within 24 hours after procedure
  Technical success is defined as post-implant dosimetry achieving D90 ≥ 90 Gy and V100 ≥ 85% without major intraoperative or immediate postoperative complications (CTCAE Grade ≥3).
Dosimetric Superiority of PET/CT-Guided Implantation | Immediately after implantation (dosimetric verification)
  Comparison of mean D90 between PET/CT-guided and CT-guided groups. Superiority is defined as a ≥10 Gy improvement in D90 or ≥5% increase in V100 coverage.
Local Control Rate at 6 Months | 6 months ± 2 weeks after implantation
  Local control is defined as complete response, partial response, or stable disease per RECIST 1.1 criteria at treated sites on follow-up imaging.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of implantation until documented disease progression or death, whichever occurs first, assessed for up to 24 months
  Time interval from treatment to progression or death, analyzed using Kaplan-Meier curves and log-rank test.
Failure-Free Survival (FFS) | From the date of implantation until the first documented treatment failure or death, assessed for up to 24 months
  Time from treatment initiation to the first occurrence of disease progression, death from any cause, treatment discontinuation due to toxicity, recurrence, or initiation of new anticancer therapy.
Overall Survival (OS) | From implantation until death from any cause, assessed for up to 24 months
  Time from implantation to death from any cause, evaluated by Kaplan-Meier method.
Pain Relief Rate | Baseline, 1, 3, and 6 months post-treatment
  Pain relief rate is defined as the proportion of patients achieving a clinically meaningful reduction in pain intensity, defined as either a ≥2-point absolute decrease or a ≥30% relative decrease from baseline, as assessed by the Visual Analogue Scale (VAS). The VAS is a 0-10 numeric pain rating scale, where 0 indicates no pain and 10 indicates the worst pain imaginable; higher scores indicate worse pain intensity.
Quality of Life (QoL) | Baseline, and 6 months
  Quality of life is assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Scores range from 0 to 100. Higher scores on functioning scales and global health status indicate better outcomes, while higher scores on symptom scales indicate worse symptoms.
Treatment-Related Adverse Events | From treatment initiation through 12 months post-treatment.
  Treatment-related adverse events will be assessed by recording the incidence, type, and severity of adverse events occurring after treatment. All adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

OTHER OUTCOMES:
Comparison of PET-GTV and CT-GTV | Pre-treatment (baseline imaging)
  Differences in tumor volume and spatial overlap between PET-defined and CT-defined GTVs, evaluated by Dice similarity coefficient and centroid distance.
Predictive Value of Baseline Tumor SUVmax on PET/CT for Treatment Outcomes | Baseline to 6 months
  To evaluate the predictive value of baseline tumor SUVmax measured on PET/CT for treatment outcomes, baseline SUVmax of the index lesion will be analyzed as a continuous predictor for 6-month local control using logistic regression and for progression-free survival (PFS) using a Cox proportional hazards regression model, with results summarized as odds ratios and hazard ratios with 95% confidence intervals.
Early Metabolic Response | 4-6 weeks post-treatment
  Change in SUVmax (ΔSUVmax) from baseline to 4-6 weeks and its predictive value for 6-month local control using ROC analysis.
Feasibility of SUV-Guided Dose Painting | Immediate post-implant verification
  Proportion of high-SUV subregions (SUVmax >5.0) achieving target D90 ≥120 Gy within organ-at-risk limits.
Correlation Between Tumor-Specific PET Tracer Uptake and Treatment Response | Baseline to 6 months
  Differences in diagnostic performance between FDG and tumor-specific PET tracers (e.g., PSMA, FAPI) are assessed by comparing lesion detectability, tumor-to-background contrast, and associations with treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Min Li, Dr., Study Director
Locations (1):
- The 960th Hospital of People's Liberation Army (PLA), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including baseline demographics, PET/CT imaging parameters (SUVmax, MTV, TLG), dosimetric results, and clinical outcomes (local control, PFS, FFS, OS), will be shared upon reasonable request after publication of the main study results. Data will be available for qualified researchers conducting methodologically sound studies related to radiomics, brachytherapy, or PET-guided radiation optimization. Requests should be submitted to the principal investigator via institutional contact email. Access will require a data sharing agreement to ensure patient privacy and compliance with institutional and ethical standards.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) will be available beginning 6 months after publication of the primary study results and will remain available for 5 years following publication, or until the main study database is closed, whichever occurs first.
Access Criteria: Qualified researchers affiliated with academic institutions or recognized research organizations may request access to de-identified individual participant data (IPD), including imaging-derived parameters, dosimetric results, and clinical outcome data. Requests must include a brief research proposal describing the scientific rationale, objectives, and planned analyses. Approval will be granted by the study's principal investigator and institutional ethics committee. Data will be shared through secure institutional data transfer systems after execution of a formal data sharing agreement that ensures patient confidentiality and compliance with applicable privacy regulations.